CLINICAL TRIAL: NCT03047629
Title: A Multi-Center, Single-Dose, Multiple-Dose, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered ENT-01 for the Treatment of Parkinson's Disease Related Constipation
Brief Title: Evaluation of Safety and Tolerability of ENT-01 for the Treatment of Parkinson's Disease Related Constipation
Acronym: RASMET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Enterin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENT-01
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Parkinson's Disease; Constipation
Keywords: non-motor symptoms
MeSH Terms: conditions — Parkinson Disease; Constipation

STUDY DESIGN:
Intervention Model Description: Phase 1 is a single group; Phase 2 will begin subsequent to the safe completion of Phase 1. Phase 2 patients will undergo randomization for parallel study during one period of observation of the course of the study phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENT-01 (Experimental): ENT-01 at a to-be-determined dose taken by mouth every day upon awakening.
  Interventions: Drug: ENT-01
- Placebo Comparator (Placebo Comparator): Placebo to be taken by mouth every day upon awakening
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ENT-01 — Daily dosing with ENT-01. ENT-01 is an orally administered proprietary substance formulated as a small 25mg coated tablet. Dosing will range from 25-200mg, and the dose will be taken upon awakening on an empty stomach with 8oz water simultaneous to dopamine.
  Arms: ENT-01
Other: Placebo — Daily dosing with a placebo
  Arms: Placebo Comparator

SUMMARY:
This is a Phase 1/2a study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of an orally-administered medication to relieve symptoms of constipation associated with Parkinson's Disease. Ten patients will be enrolled in Phase 1, and will be studied over an 8-12 week period. Forty patients will be enrolled in Phase 2, and will be studied over an 8-10 week period. All subjects will receive the study drug during one of the observational periods of the study.

DETAILED DESCRIPTION:
Phase 1 will enroll 10 patients to assess the safety, tolerability, and pharmacokinetics of single escalating doses over a 30-60 day period. The dose-escalation period will be preceded by a 2-week run in period and followed by a 2-week wash-out period.

Phase 2 follow the safe completion of Phase 1. It will enroll 40 patients and is composed of 4 periods of study: 1) a 2-week run-in period, 2) a 3-5 week escalating dose period to identify a prokinetic dose in the initial set of 10 patients, 3) a 1-week period of randomized dosing (placebo versus the previously identified pro-kinetic dose), and 4) a 2-week wash-out period. Pharmacodynamics will be assessed along with safety and tolerability. Relative outcomes will be compared within each patient and across groups for the randomized dosing period.

Frequency of bowel movements and other non-motor symptoms of Parkinson's Disease will be collected over the course of both phases.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson's disease diagnosis confirmed by a neurologist specializing in movement disorders
2. Insufficient criteria for a diagnosis of Irritable Bowel Syndrome
3. Constipation for over 6 months, unresponsive to Milk of Magnesia, and requiring at least weekly treatment using an oral laxative, stool softener, bulking agent, and/or a suppository, and dissatisfaction with current treatment.
4. Body Mass Index is 18-40 kg/m2
5. At least 2 of the Rome IV functional constipation criteria are met
6. Loose stools are rarely present without the use of laxatives
7. Patient is willing and able to sign informed consent and comply with all study procedures
8. Patients must be able to read, understand, and accurately record data into the diary to guarantee full participation in the study

   Females only:
9. Must have negative serum or urine pregnancy tests and must not be lactating
10. If of child-bearing age: Must agree to using a hormonal (i.e., oral, implantable, or injectable) and either single- or double-barrier method of birth control throughout the study period. A vasectomized partner will be allowed as one in conjunction with another single-barrier method.
11. If unable to have children: Must have this documented in the case report form (i.e., ubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone in women less than 60 years of age.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures
2. Diagnosis of secondary constipation beyond that of PD
3. Structural or metabolic diseases that affect the GI system
4. Functional GI disorder
5. Unable or unwilling to withdraw from taking the following medications 2 weeks prior to the dose-escalation period and throughout the study: Laxatives, opiates, sedatives, hypnotics, anti-histamines, protein pump inhibitors or any medications which may cause constipation
6. History of recent major surgery (within 60 days of screening)
7. Any clinically significant abnormalities on screening laboratories or physical examination as determined by the Investigator
8. Neurological disorder other than PD
9. On treatment with intra-jejunal dopamine
10. Treatment with COMT inhibitors for fewer than 4 weeks (entacapone, tolcapone, Stalevo)
11. Unable to maintain a stable diet regimen
12. Patients with a cognitive impairment that preclude them from understanding the informed consent
13. Patients placed under legal guardianship
14. Acute GI illness within 48 hours of the baseline period
15. History of major GI surgery (e.g. previous abdominal surgery, including cholecystectomy), except that patients with uncomplicated appendectomy are allowed
16. ALT or AST > 1.5 X upper limit of normal (ULN) during screening
17. Females who are pregnant or breastfeeding
18. History of excessive alcohol use or substance abuse
19. Patient or caregiver unable to administer daily oral dosing
20. Participation in an investigational clinical study within the 6 months prior to dosing in the present study
21. Any other reason, which in the opinion of the Investigator would confound proper interpretation of the study

Ages: 30 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Barbut, MD FRCP, Study Chair — Enterin Inc.; Steven Frucht, MD, Principal Investigator — NYU Langone Health; Robert Hauser, MD MBA, Principal Investigator — University of South Florida
Locations (15):
- United States (15):
  - Keck Hospital of University of Southern California, Los Angeles, California
  - Rocky Mountain Movement Disorders Center, PC, Englewood, Colorado
  - Georgetown Universtiy, Department of Neurology, Washington D.C., District of Columbia
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Neuroscience Research, University of Florida Jacksonville, Jacksonville, Florida
  - MEDSOL Clinical Research, Port Charlotte, Florida
  - Sarasota Memory Hospital Clinical Research Ctr., Sarasota, Florida
  - Suncoast Neuroscience Associates, Inc, St. Petersburg, Florida
  - USF Health Byrd Parkinson's Disease Movement Disorders Center of Excellence, Tampa, Florida
  - Quest Research Institute, Farmington Hills, Michigan
  - Movement Disorders Division, Mt. Sinai School of Medicine, New York, New York
  - Riverhills Healthcare, Inc., Cincinnati, Ohio
  - Parkinson's & Movement Disorders Center, UH Cleveland Medical Center, Cleveland, Ohio
  - Penn State Health, Department of Neurology, Hershey, Pennsylvania
  - Thomas Jefferson University, Department of Neurology, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be shared with other clinical researchers outside of this study that are involved in similar research at non-participating institutions.

REFERENCES:
- [Result] Hauser RA, Sutherland D, Madrid JA, Rol MA, Frucht S, Isaacson S, Pagan F, Maddux BN, Li G, Tse W, Walter BL, Kumar R, Kremens D, Lew MF, Ellenbogen A, Oguh O, Vasquez A, Kinney W, Lowery M, Resnick M, Huff N, Posner J, Ballman KV, Harvey BE, Camilleri M, Zasloff M, Barbut D. Targeting neurons in the gastrointestinal tract to treat Parkinson's disease. Clin Park Relat Disord. 2019 Jul 2;1:2-7. doi: 10.1016/j.prdoa.2019.06.001. eCollection 2019. PMID 34316590

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 subjects signed informed consent. 6 were screen failed during the run-in period and were not eligible to continue into the dose escalation period.
Groups:
- Stage 1: Patients will begin with a dose level of 25 mg taken daily. Patients will dose escalated until they reach a maximum dose level of 200 mg daily or experience a dose limiting toxicity.
- Stage 2: ENT-01: Patients will begin with a dose level of 75 mg taken daily. Patients will dose escalated until they reach a maximum dose level of 175 mg daily, experience a dose limiting toxicity or have a complete spontaneous bowel movement
- Stage 2: Placebo Comparator: Patients randomized to receive placebo taken by mouth every day upon awakening
Period: Overall Study
Arm/Group | Stage 1 | Stage 2: ENT-01 | Stage 2: Placebo Comparator
Started | 10 | 26 | 8
Completed | 9 | 20 | 8
Not Completed | 1 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stage 1: Sentinel group to establish safe and tolerable dose of ENT-01
  Patients will begin with a dose level of 25 mg taken daily. Patients will dose escalated until they reach a maximum dose level of 200 mg daily or experience a dose limiting toxicity.
- ENT-01: ENT-01: Daily dosing with ENT-01.
  Patients will begin with a dose level of 75 mg taken daily. Patients will dose escalated until they reach a maximum dose level of 175 mg daily, experience a dose limiting toxicity or have a complete spontaneous bowel movement
- Total: Total of all reporting groups
Arm/Group | Stage 1 | ENT-01 | Placebo Comparator | Total
Number analyzed (Participants) | 10 | 26 | 8 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (4.88) | 72.6 (7.52) | 73.1 (7.41) | 70.4 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 14
  Male | 5 | 20 | 5 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 9 | 26 | 7 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 26 | 8 | 44
Constipation Severity- Complete Spontaneous Bowel Movement per week [Count of Participants; unit: Participants]
  0-1 per week | 4 | 17 | 5 | 26
  1.1-2 per week | 4 | 7 | 2 | 13
  2.1-3 per week | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events.
Description: Specific treatment related events of recurrent vomiting, recurrent diarrhea, abdominal pain, and hypotension will be assessed with respect to grade and frequency of occurrence.
Time Frame: Through study completion, up to 11 weeks
Population: Analysis completed as stage 1 and stage 2
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2: Placebo Comparator: Placebo to be taken by mouth every day upon awakening
  Placebo: Daily dosing with a placebo
Arm/Group | Stage 1 | Stage 2: ENT-01 | Stage 2: Placebo Comparator
Number analyzed (Participants) | 10 | 24 | 8
Participants | 9 | 16 | 1

2. Secondary Outcome: Frequency of Bowel Movements
Description: The frequency of spontaneous bowel movements will be assessed at each dose across the study population and compared to baseline measures.
Time Frame: Through study completion, up to 11 weeks
Population: Frequency of bowel movements was abondoned in protocol amendment date 01 Feb 2018.
Arm/Group | Stage 2: ENT-01 | Stage 2: Placebo Comparator
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected after the start of investigational product through the end of study visit, up to 11 weeks. Serious adverse events were to be reported within 30 days of last dose of study medication
Description: NA. Adverse event collection does not differ from clinicaltrials.gov
Groups:
- Stage 1: ENT-01: Sentinel group to establish safe and tolerable dose of ENT-01
  Patients will begin with a dose level of 25 mg taken daily. Patients will dose escalated until they reach a maximum dose level of 200 mg daily or experience a dose limiting toxicity.
Arm/Group | Stage 1: ENT-01 | Stage 2: ENT-01 | Stage 2: Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/26 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/26 | 0/8
Other Adverse Events (participants affected / at risk) | 10/10 | 26/26 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: ENT-01 (N=10) | Stage 2: ENT-01 (N=26) | Stage 2: Placebo Comparator (N=8)
Abdominal Distension (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 13 | 2
Flatulance (Gastrointestinal disorders) | 2 | 1 | 0
Mucus Stools (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 14 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 5 | 1
Headache (Nervous system disorders) | 1 | 2 | 0
Loss of Appetite (Gastrointestinal disorders) | 1 | 0 | 0
Worsening Acid Reflux (Gastrointestinal disorders) | 0 | 1 | 1
Worsening Hemmorrhoid (Gastrointestinal disorders) | 0 | 0 | 0
Lower GI bleed (Gastrointestinal disorders) | 0 | 1 | 0
Blood in Urine (Renal and urinary disorders) | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1
Urinary Tract Infection (Renal and urinary disorders) | 0 | 3 | 0
Increased Urinary frequency (Renal and urinary disorders) | 0 | 2 | 0
Skin lesions- rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Eye Infection (Eye disorders) | 0 | 1 | 0
Difficulty falling asleep (General disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT03047629/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03047629/SAP_001.pdf